CLINICAL TRIAL: NCT00467922
Title: A Randomized Prospective Double Blind Assessment of Goal-Directed Intraoperative Fluid Management in Hand Assisted Laparoscopic Colectomy: Standard Care Versus Either Colloid and Crystalloid
Brief Title: An Assessment of Goal-Directed Intraoperative Fluid Management in Hand Assisted Laparoscopic Colectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Corewell Health West (Other)
Collaborators: Deltex Medical, Inc. (Industry)
Responsible Party: Dr. Anthony Senagore, Spectrum Health
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2007-109; 2007-109
Record Dates: First submitted 2007-04-27; First posted 2007-05-01 (Estimated); Last update posted 2009-10-21 (Estimated); Status verified 2009-10

CONDITIONS: Crohn's Disease; Ulcerative Colitis; Rectal Cancer; Colon Cancer; Colon Polyps; Rectal Polyps; Diverticulitis
Keywords: Hand-assisted colorectal surgery; colorectal disease; Crohn's; diverticulitis; Colorectal resections
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Rectal Neoplasms; Colonic Neoplasms; Colonic Polyps; Diverticulitis | interventions — Hydroxyethyl Starch Derivatives; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Hextend — Assessment of Goal-Directed Intraoperative Fluid Management in Hand Assisted Laparoscopic Colectomy: Standard Care versus Either Colloid and Crystalloid
Drug: Lactated Ringers — Assessment of Goal-Directed Intraoperative Fluid Management in Hand Assisted Laparoscopic Colectomy: Standard Care versus Either Colloid and Crystalloid

SUMMARY:
The purpose of this study is to find out if guided fluid administration with the esophageal monitor is superior to standard fluid administration and whether use of the hetastarch or lactated ringers offers different benefits with respect to length of stay in the hospital after hand-assisted colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnoses of Crohn's disease, ulcerative colitis, rectal or colon cancer, colon or rectal polyps and chronic or subacute diverticulitis
2. Subjects who will undergo hand-assisted laparoscopic colectomy for benign or malignant pathology

Exclusion Criteria:

1. Patients requiring stoma formation as part of the operative procedure
2. Patients undergoing loop ileostomy or colostomy closure thru the stomal site
3. Bowel obstruction, coagulopathy, significant renal or hepatic dysfunction (creatinine >1.6 or liver enzymes > 50% upper limit of normal values)
4. Congestive heart failure, unstable angina, or valvular heart disease with New York Heart Classification >2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Determine the relative effects of a standard, colloid or crystalloid based strategy for hand-assisted laparoscopic colectomy surgery on decreasing length of stay | 90 days

SECONDARY OUTCOMES:
1. Determine the effects of the three fluid management strategies on post-operative fluid requirements in colorectal surgery. on the incidence and severity of post-operative complications. on return of gastrointestinal function. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Senagore, MD, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health, Grand Rapids, Michigan, United States